CLINICAL TRIAL: NCT04711590
Title: Association Between Change of Microcirculation After Spontaneous Breathing Trial and Ventilator Weaning
Brief Title: Microcirculation in Spontaneous Breathing Trial
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201909036RINB
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-04

CONDITIONS: Critically Ill
Keywords: ventilator; weaning; microcirculation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful extubation: The patients pass the spontaneous breathing trial and are successful extubated without reintubation within 72 hours. .
  Interventions: Other: Microcirculation examination
- Failed extubation: The patients pass the spontaneous breathing trial and are successful extubated with reintubation within 72 hours. .
  Interventions: Other: Microcirculation examination

INTERVENTIONS:
Other: Microcirculation examination — Sublingual microcirculation images were recorded using an incident dark-field video microscope

SUMMARY:
Weaning ventilator support in critically ill patients is crucial. Both delayed extubation and unexpected early reintubation are harmful to the patients. Weaning parameters and spontaneous breathing trial are used to investigate the indication and predict the successful extubation. Hemodynamic stability and physical reserve are important indicators as well. Microcirculation parameters are known to be more sensitive to the change of hemodynamic status than macrocirculation parameters. We hypothesize that the change of sublingual microcirculation before and after spontaneous breathing trial is different between the the patients with successful extubation and the patients with failed extubation. Thus, this study measures sublingual microcirculation in patients receiving spontaneous breathing trial and record the extubation status (successful or failed). The microcirculation parameters before and after spontaneous breathing trial are compared between the the patients with successful extubation and the patients with failed extubation.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients received ventilator longer than 12 hours
* ready for spontaneous breathing trial
* GCS coma score equal or higher than 8

Exclusion Criteria:

* aged less than 20 years
* patient with tracheostomy
* patient and patients' relatives are non-native speakers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients who are ready for weaning ventilator support and receive spontaneous breathing trial.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Initial total vessel density | 0 hour
  Total vessel density measured by Cytocam before and after spontaneous breathing trial
Change of total vessel density | baseline and 1 hour
  The difference between the total vessel density measure by Cytocam before and after spontaneous breathing trial

SECONDARY OUTCOMES:
Initial perfused vessel density | 0 hour
  Perfused vessel density measured by Cytocam before spontaneous breathing trial
Change of perfused vessel density | baseline and 1 hour
  The difference between the perfused vessel density measure by Cytocam before and after spontaneous breathing trial

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study will be available from the corresponding author upon reasonable request and approval of the research ethic committee.